CLINICAL TRIAL: NCT04587856
Title: Molecular Mechanisms of Disease Relapse After Allogenic Stem Cell Transplantation in Patients With Myelodysplastic Syndrome
Brief Title: Molecular Mechanisms of Disease Relapse After Allogenic Stem Cell Transplantation in MDS Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MDS0620
Record Dates: First submitted 2020-09-24; First posted 2020-10-14 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological evaluation (Other): evaluation of molecular changes in CD34+ blast cells at the time of relapse after allo-HSCT.
  Interventions: Other: bone marrow withdrawal

INTERVENTIONS:
Other: bone marrow withdrawal — bone marrow samples evaluation

SUMMARY:
This is a biological study for adult MDS patients who undergo HSCT procedure. Viable bone marrow samples will be collected and cryopreserved from MDS patients before transplantation and at clinical disease recurrence. CD34+ blast cells at disease relapse after HSCT will be compared with CD34+ cells collected before transplant to study genomic and transcriptomic changes.

DETAILED DESCRIPTION:
This is a biological study for adult MDS patients who undergo HSCT procedure.The research is focused on the study of biological mechanisms of disease relapse after HSCT in MDS to provide the rationale to develop pre-emptive strategies in patients with high risk of transplant failure.

Viable bone marrow samples will be collected and cryopreserved from MDS patients before transplantation and at clinical disease recurrence.

CD34+ blast cells at disease relapse after HSCT will be compared with CD34+ cells collected before transplant by using Single-cell sequencing.

To study genomic and transcriptomic changes in CD34+ blast cells at disease relapse after HSCT will be used TARGET-seq in parallel with unbiased whole-transcriptome analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS according to 2016 WHO criteria
* Aged 18y or older
* Patients who will receive allogeneic stem cell transplantation (HSCT)
* Signed written informed consent according to ICH/EU/GCP and national local laws

Exclusion Criteria:

* Second HSCT procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
CD34+ blast cells modifications | at 24 months
  Difference in frequency distribution of CD34+ blast cells mutations between transplant and relapse.

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Unità di Ricerca e di Malattie del sangue - Ematologia S. Luca Vecchio, Florence
  - AOU San Martino-IST-Ematologia 1, Genova
  - Sezione di Ematologia - Ospedale S.Maria della Misericordia, Perugia
  - Dip. di Medicina Trasl. E di Precisione - U.O.C. Ematologia, Roma
  - Policlinico Tor Vergata, Roma
  - Ististuto Clinico Humanitas - Rozzano - Uo Oncologia Medica Ed Ematologia, Rozzano